CLINICAL TRIAL: NCT05242094
Title: Assessment of Depressive and Anxiety Symptoms in Post-COVID-19 Patients During In-Hospital Pulmonary Reha-bilitation With Support of Virtual Reality
Brief Title: Pulmonary Rehabilitation Implemented With VR for Post-COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID_1
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: COVID-19; Pulmonary rehabilitation; Virtual Reality
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Traditional Pulmonary Rehabilitation
  Interventions: Procedure: Pulmonary Rehabilitation Program
- Group 2 (Experimental): Pulmonary Rehabilitation in Virtual Reality
  Interventions: Procedure: Pulmonary Rehabilitation Program

INTERVENTIONS:
Procedure: Pulmonary Rehabilitation Program — An in-patients 3-week high intensity rehabilitation program, five times a week, was used as the intervention treatment. The author's pulmonary rehabilitation program was programmed based on previous experience in patients with COPD. A holistic pulmonary rehabilitation program with combined treatment focused on increasing exercise capacity, restoring lung function, and supporting mental health, developed by a multidisciplinary team, was introduced. Based on the patient's submaximal exercise tolerance test results, the qualification for one of the respiratory physiotherapy models differing in therapy intensity was performed. Rehabilitation models included exercise capacity training on a cycle ergometer, breathing exercises, general fitness exercises, resistance training, and relaxation.

SUMMARY:
Although the COVID-19 pandemic was announced almost 2 years ago, societies are still facing the effects not only of individuals but also of entire populations. Clinical symptoms in patients depending on the variant of the virus range from fever, sore throat, cough, fatigue, or gastrointestinal or neurological symptoms. Symptoms of respiratory failure also occur, as well as heart and kidney damage. Therefore, it is important to implement appropriate pulmonary rehabilitation programs to counteract the effects of the disease. The current project aims to evaluate the effectiveness of a comprehensive pulmonary rehabilitation program for patients hospitalized for SARS-CoV2 infection.

DETAILED DESCRIPTION:
Initial studies indicated that approximately 60 days after the first COVID-19 symptom onset, only 13% of patients previously hospitalized for COVID-19 were reported to be essentially free of any COVID-19-related symptoms, while 32% had one or two symptoms and 55% had three or more symptoms. Furthermore, the COVID-19 pandemic gives rise to new psychosocial and emotional stressors for recovering patients, including social isolation, physical distancing, loss of employment and uncertainties about the future. In the confrontation of such an uncertain prognosis, it seems justified to introduce preventive actions against the development of pandemic-related adverse effects. To date, only few publications assessed the effectiveness of early post-hospital rehabilitation of patients with COVID-19. This project is aimed to propose an innovative comprehensive intervention based on a stationary pulmonary rehabilitation (PR) programme for COVID-19 survivors. Moreover, this project assumes the use of virtual reality (VR) in rehabilitation processes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals hospitalized for COVID-19.

Exclusion Criteria:

* Failure to consent to participate in research,
* pneumonia,
* evidence of ischemic heart disease/acute changes on ECG,
* uncontrolled hypertension,
* insulin dependent diabetes mellitus,
* inability to exercise independently or musculoskeletal/neurological conditions that would prevent completion of the course,
* lung cancer,
* cognitive disorders, or Mini-Mental State Examination < 24.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 10 minutes
  The Polish version of the Hospital Anxiety and Depression Scale (HADS) was used to assess depression and anxiety in patients. The questionnaire is considered a reliable method of assessing anxiety and depression [15]. The HADS questionnaire consists of 14 questions scored on a 4-point (0 to 3) scale.
Functional Capacity | 20 minutes
  Functional capacity assessment included exercise capacity (6-minute walk test) and lung ventilation function (spirometry).

CONTACTS AND LOCATIONS:
Locations (1):
- MSWiA Specialist Hospital in Głuchołazy, Głuchołazy, Opole Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Data will not be available.